CLINICAL TRIAL: NCT06700902
Title: A Randomized Controlled Trial of Taking Action Planning for College Students With Serious Mental Illnesses
Brief Title: Taking Action for College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 31680
Record Dates: First submitted 2024-08-30; First posted 2024-11-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Schizophrenia
Keywords: Taking Action; Recovery; Wellness; Serious Mental Illness; College Students
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Intervention Model Description: A total of 60 students will be enrolled in the study per semester, 30 of whom will be randomized to Taking Action and 30 to the control condition. Enrollment will occur over a period of 5 semesters, with two Taking Action groups running concurrently each semester. Randomization will occur at the participant-level and will be facilitated by using an HIPAA-compliant, Internet-based randomization service (studyrandomizer.com). The research assistant, who will be blind to the random allocation sequence, will enter participants into the randomization service after completion of the baseline interview and notify them of the condition to which they are assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taking Action Intervention Condition (Experimental): Participants in the experimental condition will participate in the Taking Action intervention.
  Interventions: Behavioral: Taking Action
- Information Only Control Condition (No Intervention): Participants in the information only control condition will not participate in any intervention but will be given access to a resource entitled, "A Practical Guide for People with Disabilities Who Want to Go to College".

INTERVENTIONS:
Behavioral: Taking Action — Participants in the experimental condition will participate in the Taking Action intervention, which will be delivered in a small group format in 5 weekly 2.5 hour videoconferencing sessions. Taking Action will be implemented using materials available on SAMHSA's website (https://www.co.ozaukee.wi.us/DocumentCenter/View/8198/Taking-Action-A-MH-Recovery-Self-Help-Ed-Program?bidId=). The process will include an overview of key recovery and wellness concepts and the development of an individualized wellness toolbox, which is a list of skills and strategies that a person already uses or would like to use to maintain or regain wellness. Then, participants will make plans for monitoring and addressing distressing mental health symptoms. Instructional techniques will include lectures, discussions, personal examples from facilitators and participants own lives to illustrate key concepts related to self-management, individual and group exercises, and voluntary action plans between meetings.
  Arms: Taking Action Intervention Condition

SUMMARY:
The goal of this research is to investigate whether a peer-delivered illness self-management program called Taking Action can help college students with serious mental illnesses. Participants will be randomly assigned to either the experimental condition (Taking Action) or the control condition (information only). Participants in the experimental condition will attend five 2.5-hour Taking Action sessions. Participants will complete three interviews (baseline, post-intervention, and follow-up) to assess how well the program works, is liked, and benefits students clinically and academically. The investigators seek to test the following hypotheses: Compared to controls, students who do the Taking Action program will report greater improvements in mental health self-management attitudes, skills, and behaviors and will report greater improvements in mental health symptoms and recovery, and better academic outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility, acceptability, and effectiveness associated with Taking Action for college students with serious mental illnesses (SMI). The study will be a randomized controlled trial. The investigators plan to recruit 300 college students with SMI to participate in the study. A total of 60 students will be enrolled in the study per semester, 30 of whom will be randomized to Taking Action and 30 to the control condition. Enrollment will occur over a period of 5 semesters, with two Taking Action groups running concurrently each semester. The investigators will recruit from within Temple University and other colleges and universities in the United States.

Participants will be randomly assigned to one of two groups, the experimental condition (Taking Action) or the control condition (information only). Participants in the experimental condition will attend five 2.5-hour Taking Action sessions that will be delivered in a small group format online via videoconferencing.

All participants will complete 3 research interviews: baseline, post-intervention and follow-up, lasting about 1.5 hours each. Data related to the feasibility of research and intervention procedures, acceptability of the intervention, and clinical and academic outcomes will be collected and analyzed. The investigators will assess the feasibility of the intervention procedures by tracking data pertaining to recruitment, retention, and assessment using CONSORT guidelines, and data related to implementation of the intervention (i.e., fidelity, number of intervention meetings attended by participant). Fidelity to Taking Action will be assessed using a facilitator checklist based on prescribed content, procedures, and materials for each Taking Action session. Facilitators will also maintain attendance logs in RedCAP for each Taking Action session. The investigators will assess the acceptability of the intervention via quantitative and qualitative questions administered at post-intervention about participants' level of satisfaction and experiences with the intervention. The investigators will assess the clinical and academic outcomes of the intervention using the Mechanisms of Action Scale, Hopkins Symptom Checklist, Recovery Assessment Scale, College Persistence Questionnaire, Perceived Competence Scale, College Self-Efficacy Inventory, Study Habits Inventory, and Procrastination Assessment Scale - Students. Some exploratory measures will also be included in the interviews.

Feasibility and quantitative acceptability data will be reported using descriptive statistics. Qualitative acceptability data will be analyzed using thematic analysis. To examine the impact of Taking Action on mental health and academic outcomes random effect ANOVAs on repeated measures data in PROC MIXES (SAS) will be used to compare the experimental and control groups over time on the various measures. Prior to running the random effects ANOVAs above, the investigators will examine whether the experimental and control groups were different at baseline on any background characteristics despite randomization, and if so, control for them in the analyses. In addition, exploratory analyses will be conducted to provide insight regarding the characteristics of students who are most likely to benefit from Taking Action.

The investigators will recruit 300 individuals, which, with an estimated attrition rate of 25% based on previous experience with this population, will yield a sample of 225 participants with complete data. In a repeated measures ANOVA with two groups, three time points, and the correlation between repeated measures assumed to be 0.5, the investigators will be able to achieve .80 power to detect a small effect size of f=.085 in a time*group interaction term when the probability of a type I error, alpha, is set at .05. Even so, the investigators anticipate these power estimates are conservative, because of the use of PROC MIXED in SAS for analyzing repeated measures data. PROC MIXED does not discard participants with missing data at some time points, making the impact of missing data and attrition on power much less severe. GPower was used for power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a 2- or 4-year postsecondary educational institution in the United States (and are able to present a valid student ID card)
* Experiencing a serious mental illness, as operationalized by either:
* A score of 13 or higher on the K-6 Screening Scale for serious mental illness
* Self-reported psychiatric diagnosis of schizophrenia-spectrum or major affective disorder and self-reported lifetime functional impairment due to experiencing mental health challenges
* 18 years of age or older
* Have consistent access to a computer or smartphone and the Internet for communications
* No prior WRAP or Taking Action education

Exclusion Criteria:

* Expected to graduate or complete their program within 2 semesters
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline in Mental Health Symptoms | Baseline, Immediately After the Intervention, and 3-Month Follow-Up
  The Brief Symptom Inventory is a validated instrument used to assess mental health symptoms. The mean T-score is 50, with higher scores indicating worse outcome.
  Change = (3-Month Follow-Up Score - Baseline Score).
Changes from Baseline in Perceived Recovery | Baseline, Immediately After the Intervention, and 3-Month Follow-Up
  The Recovery Assessment Scale is a validated instrument used to assess perceived recovery from mental illness. Scores range from 1 to 5 with higher scores indicating greater perceived recovery.
  Change = (3-Month Follow-Up Score - Baseline Score).

SECONDARY OUTCOMES:
Changes from Baseline in Intention to Persist in College | Baseline, Immediately After the Intervention, and 3-Month Follow-Up
  The College Persistence Questionnaire is a validated instrument used to assess intention to persist in school. Scores range from -16 to +16 with higher scores indicating greater intention to persist in school.
  Change = (3-Month Follow-Up Score - Baseline Score).
Changes from Baseline in Perceived Competence in Educational Environment | Baseline, Immediately After the Intervention, and 3-Month Follow-Up
  The Perceived Competence Scale is a validated instrument used to assess perceived competence that will be applied to an educational environment by asking how true items are "with respect to your learning in your school courses." Scores range from 1-7, with higher scores indicating greater perceived competence.
  Change = (3-Month Follow-Up Score - Baseline Score).
Changes from Baseline in Study Habits | Baseline, Immediately After the Intervention, and 3-Month Follow-Up
  The Study Habits Inventory is a validated instrument used to assess study habits. Scores range from 1 to 7 with higher scores indicating better study habits.
  Change = (3-Month Follow-Up Score - Baseline Score).
Changes from Baseline in Procrastination | Baseline, Immediately After the Intervention, and 3-Month Follow-Up
  The Procrastination Assessment Scale - Students is a validated measure used assess procrastination. Scores range from 1 to 5 with higher scores indicating greater procrastination.
  Change = (3-Month Follow-Up Score - Baseline Score).
Change from Baseline in College Self-Efficacy | Baseline, Immediately After the Intervention, 3 Month Follow-Up
  The College Self-Efficacy Inventory is a validated measure that assesses perceived self-efficacy in a college context. Scores range from 1 to 10 with higher scores indicating a better outcome. Change = (3-Month Follow-Up Score - Baseline Score).

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No